CLINICAL TRIAL: NCT01903226
Title: High Intensity Aerobic Training in Persons With Incomplete Spinal Cord Injury
Brief Title: Intervention Study to Assess the Effects of Moderate and High Intensity Aerobic Training on Physical Capacity and Activity Level in Persons With Incomplete Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Matthijs Ferdinand Wouda, PhD candidate, Sunnaas Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPREK
Record Dates: First submitted 2013-07-10; First posted 2013-07-19 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; physical capacity; energy expenditure; training
MeSH Terms: conditions — Spinal Cord Injuries | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High intensity training (Experimental): Patients in this group will perform high aerobic intensity training, in 30 minutes, twice a week, in a 12 week period.
  Interventions: Other: High intensity training
- Moderate intensity training (Experimental): Patients in this group will perform moderate aerobic intensity training, in 45 minutes, three times a week, in a 12 week period.
  Interventions: Other: Moderate intensity training
- controll (No Intervention): Patients in this group will perform no (additional) training.

INTERVENTIONS:
Other: High intensity training
  Arms: High intensity training
Other: Moderate intensity training
  Arms: Moderate intensity training

SUMMARY:
The aims of this study are to assess the effects of medium versus high intensity 12-week adjusted training programs on physical capacity in persons with incomplete SCI, early after discharge from primary rehabilitation, and to investigate if the training program induces a more active lifestyle in terms of increased daily energy expenditure.

DETAILED DESCRIPTION:
Design:

Randomized controlled trial.

Participants:

45 subjects, between 18 and 65 years of age, will be recruited with the following inclusion criteria: Traumatic spinal cord injury, incomplete lesions (classified as ASIA D), admitted to Sunnaas Rehabilitation Hospital for primary rehabilitation, and able to walk for 5 minutes on the treadmill (without assistive aids) at 4 km/hour.

Subjects with cardiovascular diseases, progressive diseases and severe psychiatric conditions will be excluded.

Procedures:

The participants will be included after medical approval (by a specialist in physical medicine and rehabilitation) and before being discharged from primary rehabilitation. During the last week at the hospital, usually between 3 to 6 months post injury, a pre-test to examine physical capacity will be performed; maximal exercise test on a treadmill and six-minute walking test (Fig. 1).

After the pre-test the participants will be randomized into one of three groups; Intervention Group I (high intensity training), Intervention Group II (medium intensity training), and a Control Group (treatment as usual, no additional training). To achieve balanced randomization (the compared groups should have about the same size), we will use block randomization. A computer random number generator will be used, with a block size of 15 and an allocation ratio of 1:1.

The subjects in the training groups will have practical training at the hospital in how to perform moderate or high intensity training. They will be taught how to apply a heart rate monitor and how to use it during training sessions.

At discharge from primary rehabilitation, and before start-up of the 12 week training program, the physical activity level (energy expenditure; kilo joule (kJ) · min -1) will be monitored by wearing a SWA for seven days in the home situation.

After having completed the training program, the participants (including those in the control group) will wear the SWA in 7 days and return to Sunnaas Rehabilitation Hospital to repeat the physical capacity tests (post-test). This procedure will also be repeated at a follow-up one year after discharge from primary rehabilitation (12-months follow-up).

All tests are performed under supervision of a physiotherapist, who has several years of experience in exercise testing. This physiotherapist is unaware of which of the three groups the patient the patient is recruited from (blind controlled trail).

Interventions:

Subjects in the two intervention groups will perform a 12 week individual training program, where 15 subjects will perform high intensity training and 15 subjects will perform a training program with moderate intensity training. Since literature indicates that SCI patients, on group level, do not improve their physical capacity after being discharged, our subjects will perform the training program in their home situation. To verify the intensity level during the training session, the participants have to wear a heart rate monitor. The heart rate will be stored for later analyses. Subjects in both training groups will be contacted, by telephone, during the first and the sixth week of the training program, to evaluate the training. A training log will be filled out by all the subjects (including those in the control group) during week 2-13.

When comparing two training programs, one must be sure that the total amount of energy expended (total oxygen uptake) is equal. The calculation of the total oxygen uptake for the different training programs is based on the relationship between %HRmax and %VO2max, established by the American College of Sports Medicine (ACSM).

Intervention group I - High intensity training The training program with high intensity will consist of two high intensity training sessions per week, using a treadmill or by outdoor walking/running. During these sessions the subjects will walk/run 4 times 4 minutes at an intensity of 85-95% of HRmax (interval training). Between the intervals, the subjects will have an active resting period (3 minutes), in which they walk at an intensity of 70% of HRmax. The subjects are free to choose which days of the week they conduct the training sessions, however, they must have at least one (resting) day in between.

Intervention group II - Moderate intensity training The training program with moderate intensity will consist of three moderate intensity training sessions per week, using a treadmill or by walking outdoor. During these sessions the subjects will walk for 45 minutes at 70% of HRmax. The subjects are free to choose which days of the week they conduct their training session Control group The subjects in the control group (n=15) will have no additional training program, but left with treatment as usual. They will, however, be offered an individual training program after the one year follow-up test.

Outcome measures

Primary outcome measures:

- Difference in VO2peak (change between pre-test and post-test 1) for both interventions groups and the control group.

Healthy, untrained subjects show about 0.5 % increase in VO2peak for every (high intensity) training session. Assuming that persons with incomplete SCI show the same increase, we need about 15 subjects to detect a mean difference of 12 % in VO2peak. Sample size calculation is based on a standard deviation of 10 % with a significance level of 0.05 and power output of 80%.

Secondary outcome measures:

* Difference in VO2peak between intervention group 1 (high intensity) and 2 (moderate intensity), after having completed the training program (post-test 1)
* Changes in VO2peak (changes between pre-test, post-test 1 and post-test 2) for both interventions groups and the control group.
* Difference in VO2peak between intervention group I (high intensity) and II (moderate intensity), one year after discharge (post-test 2).
* Difference in daily energy expenditure (kilo joule (kJ) · min -1) between pre-test, posttest 1 and post-test 2
* Difference in daily energy expenditure (kilo joule (kJ) · min -1) between intervention group I (high intensity) and II (moderate intensity), one year after discharge (post-test 2).

Data analyses and statistics:

Oxygen uptake during the last 30 seconds of the maximal exercise test will be used to estimate peak oxygen uptake (VO2peak). VO2peak of pre- and post test (1, 2 and 3) will be compared to evaluate a possible training effect. From the SWA data, the daily energy expenditure (energy expended during one week divided by 7 days) before the training program, after the training program and one year after discharge, will be compared to evaluate a possible effect of the training programs on the subjects' physical activity level.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury
* incomplete lesion (classified as ASIA D)
* admitted to Sunnaas Rehabilitation Hospital for primary rehabilitation,
* able to walk for 5 minutes on the treadmill (without assistive aids) at 4 km/hour

Exclusion Criteria:

* cardiovascular diseases
* progressive diseases
* severe psychiatric conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2017-01 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
change in VO2peak | 0 months, 3 months and 12 months
  Physical capacity (VO2peak) will be measured before intervention (baseline), after 3 months and after 1 year (12 months. Changes (from baseline) in VO2peak after 3 months and after one year is the primary outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnaas Rehabilitation Hospital, Nesoddtangen, Norway